CLINICAL TRIAL: NCT03070444
Title: Vacuum-formed Retainer Versus Bonded Retainer to Prevent Relapse After Orthodontic Treatment - A Randomized Controlled Trial About Stability and Patients' Perceptions
Brief Title: Vacuum-formed Retainer Versus Bonded Retainer to Prevent Relapse After Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Gävleborg (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFUG-557411
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Orthodontics; Retention
Keywords: Essix retainer; Vacuum-formed retainer; Cuspid-to-cuspid retainer
MeSH Terms: interventions — Orthodontic Appliances, Fixed; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: CTC retainer + Essix retainer (Experimental): The CTC is bonded directly after debonding. The Essix retainer maxilla is handed out to the patient the same day after removal of fixed appliances.
  Alginate impressions are taken at the follow-up visits. Questionnaires are completed at the follow-up visits.
  Interventions: Device: CTC retainer; Device: Essix retainer maxilla; Procedure: Alginate impression; Other: Questionnaire
- Group B: Essix retainer + Essix retainer (Active Comparator): The Essix retainer maxilla and Essix retainer mandible are handed out to the patient the same day after removal of fixed appliances.
  Alginate impressions are taken at the follow-up visits. Questionnaires are completed at the follow-up visits.
  Interventions: Device: Essix retainer maxilla; Device: Essix retainer mandible; Procedure: Alginate impression; Other: Questionnaire

INTERVENTIONS:
Device: CTC retainer — The CTC retainer consists of 0.8 hard Remanium® wire (Dentaurum, Germany) and is bonded with Tetric Flow (Ivoclar Vivadent, Liechtenstein) to the lower canines directly after debonding.
  Other Names: Fixed retainer; Bonded retainer
  Arms: Group A: CTC retainer + Essix retainer
Device: Essix retainer maxilla — The Essix retainer is made of 1 mm Essix C+® Plastic (Dentsply, USA) and is handed out to the patient the same day after removal of fixed appliances.
  Other Names: Removable retainer; Vacuum-formed retainer
Device: Essix retainer mandible — The Essix retainer is made of 1 mm Essix C+® Plastic (Dentsply, USA) and is handed out to the patient the same day after removal of fixed appliances.
  Other Names: Removable retainer; Vacuum-formed retainer
  Arms: Group B: Essix retainer + Essix retainer
Procedure: Alginate impression — Alginate impressions are taken to made the cuspid-to-cuspid and Essix retainers, respectively. Dental casts are obtained at the debond appointment and at the follow-up visits after 6, 18 and 60 months.
Other: Questionnaire — A questionnaire is completed at the follow-up visits.

SUMMARY:
The purpose of this trial is to evaluate and compare stability after orthodontic treatment with an Essix retainer and a bonded cuspid-to-cuspid retainer (CTC), respectively in the mandibular arch and longitudinally follow these patients over time up to 5 years. The patients' perceptions of the two methods are also evaluated with questionnaires during the follow-up period.

A further aim of this study is to analyze the relationship between diagnosis, treatment outcome, treatment time, age at start of treatment and stability with an Essix retainer in the maxilla.

The null hypotheses are:

* that there is no difference in retention capacity between Essix retainer and cuspid-to-cuspid retainer
* that there is no difference in patients' perception between Essix retainer and cuspid-to-cuspid retainer
* that there is no difference in retention capacity for Essix retainer in the maxilla concerning diagnosis before treatment, treatment outcomes, treatment time and age at start of treatment

DETAILED DESCRIPTION:
The study is conducted at the Orthodontic Clinic, Gävle, Sweden and consists of 104 patients. All patients are treated with fixed appliances in the upper and lower jaw (standard .022 straight wire), both with and without extractions. The patients are randomized into two groups with 52 patients in each group (Group A: cuspid-to-cuspid retainer, Group B: Essix retainer).

Dental cast are obtained at the debond appointment (T1) and at the follow-up controls after six months (T2), 18 months (T3) and 60 months (T4) for both groups.

At the visit two weeks in retention and at the follow-up visits after 6, 18 and 60 months the patients assess questionnaires in order to evaluate their experience of retention with the retention device.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with fixed appliances in both the maxilla and the mandible

Exclusion Criteria:

* Rapid Maxillary Expansion (RME) for patients with severe transversal malocclusion
* Treatment with segmented appliances
* Patients with craniofacial anomalies and patients requiring orthognatic surgery
* Patients with missing mandibular incisor

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-11-12 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anke Krämer, DDS, Principal Investigator — Folktandvården Gävleborg AB, Specialisttandvården ortdonti

IPD SHARING:
Plan to Share IPD: No
The participant data will be shared on reasonable request.

REFERENCES:
- [Background] Atack N, Harradine N, Sandy JR, Ireland AJ. Which way forward? Fixed or removable lower retainers. Angle Orthod. 2007 Nov;77(6):954-9. doi: 10.2319/103106-449.1. PMID 18004927
- [Background] Bennett ME, Tulloch JF. Understanding orthodontic treatment satisfaction from the patients' perspective: a qualitative approach. Clin Orthod Res. 1999 May;2(2):53-61. doi: 10.1111/ocr.1999.2.2.53. PMID 10534980
- [Background] Feldmann I, List T, John MT, Bondemark L. Reliability of a questionnaire assessing experiences of adolescents in orthodontic treatment. Angle Orthod. 2007 Mar;77(2):311-7. doi: 10.2319/0003-3219(2007)077[0311:ROAQAE]2.0.CO;2. PMID 17319767
- [Background] Feldmann I, List T, Bondemark L. Orthodontic anchoring techniques and its influence on pain, discomfort, and jaw function--a randomized controlled trial. Eur J Orthod. 2012 Feb;34(1):102-8. doi: 10.1093/ejo/cjq171. Epub 2011 Feb 7. PMID 21300723
- [Background] Hichens L, Rowland H, Williams A, Hollinghurst S, Ewings P, Clark S, Ireland A, Sandy J. Cost-effectiveness and patient satisfaction: Hawley and vacuum-formed retainers. Eur J Orthod. 2007 Aug;29(4):372-8. doi: 10.1093/ejo/cjm039. PMID 17702797
- [Background] Jaderberg S, Feldmann I, Engstrom C. Removable thermoplastic appliances as orthodontic retainers--a prospective study of different wear regimens. Eur J Orthod. 2012 Aug;34(4):475-9. doi: 10.1093/ejo/cjr040. Epub 2011 Apr 20. PMID 21508267
- [Background] Lindauer SJ, Shoff RC. Comparison of Essix and Hawley retainers. J Clin Orthod. 1998 Feb;32(2):95-7. No abstract available. PMID 9709631
- [Background] Littlewood SJ, Millett DT, Doubleday B, Bearn DR, Worthington HV. Retention procedures for stabilising tooth position after treatment with orthodontic braces. Cochrane Database Syst Rev. 2016 Jan 29;2016(1):CD002283. doi: 10.1002/14651858.CD002283.pub4. PMID 26824885
- [Background] Kumar AG, Bansal A. Effectiveness and acceptability of Essix and Begg retainers: a prospective study. Aust Orthod J. 2011 May;27(1):52-6. PMID 21696115
- [Background] Reitan K. Clinical and histologic observations on tooth movement during and after orthodontic treatment. Am J Orthod. 1967 Oct;53(10):721-45. doi: 10.1016/0002-9416(67)90118-2. No abstract available. PMID 5233926
- [Background] Renkema AM, Al-Assad S, Bronkhorst E, Weindel S, Katsaros C, Lisson JA. Effectiveness of lingual retainers bonded to the canines in preventing mandibular incisor relapse. Am J Orthod Dentofacial Orthop. 2008 Aug;134(2):179e1-8. doi: 10.1016/j.ajodo.2008.06.003. PMID 18675196
- [Background] Rowland H, Hichens L, Williams A, Hills D, Killingback N, Ewings P, Clark S, Ireland AJ, Sandy JR. The effectiveness of Hawley and vacuum-formed retainers: a single-center randomized controlled trial. Am J Orthod Dentofacial Orthop. 2007 Dec;132(6):730-7. doi: 10.1016/j.ajodo.2006.06.019. PMID 18068589
- [Background] Sheridan JJ, LeDoux W, McMinn R. Essix retainers: fabrication and supervision for permanent retention. J Clin Orthod. 1993 Jan;27(1):37-45. No abstract available. PMID 8478438
- [Background] Thickett E, Power S. A randomized clinical trial of thermoplastic retainer wear. Eur J Orthod. 2010 Feb;32(1):1-5. doi: 10.1093/ejo/cjp061. Epub 2009 Oct 14. PMID 19828592
- [Background] Yu Y, Sun J, Lai W, Wu T, Koshy S, Shi Z. Interventions for managing relapse of the lower front teeth after orthodontic treatment. Cochrane Database Syst Rev. 2013 Sep 6;2013(9):CD008734. doi: 10.1002/14651858.CD008734.pub2. PMID 24014170
- [Derived] Steegmans PAJ, Cavagnetto D, Reynders RAM. Which orthodontic retention protocol should I implement? A critical assessment of a randomised controlled trial. Evid Based Dent. 2022 Dec;23(4):162-165. doi: 10.1038/s41432-022-0845-7. Epub 2022 Dec 16. PMID 36526846
- [Derived] Kramer A, Sjostrom M, Apelthun C, Hallman M, Feldmann I. Post-treatment stability after 5 years of retention with vacuum-formed and bonded retainers-a randomized controlled trial. Eur J Orthod. 2023 Feb 10;45(1):68-78. doi: 10.1093/ejo/cjac043. PMID 35968668
- [Derived] Kramer A, Sjostrom M, Hallman M, Feldmann I. Vacuum-formed retainers and bonded retainers for dental stabilization-a randomized controlled trial. Part II: patients' perceptions 6 and 18 months after orthodontic treatment. Eur J Orthod. 2021 Apr 3;43(2):136-143. doi: 10.1093/ejo/cjaa039. PMID 32613244
- [Derived] Kramer A, Sjostrom M, Hallman M, Feldmann I. Vacuum-formed retainer versus bonded retainer for dental stabilization in the mandible-a randomized controlled trial. Part I: retentive capacity 6 and 18 months after orthodontic treatment. Eur J Orthod. 2020 Nov 3;42(5):551-558. doi: 10.1093/ejo/cjz072. PMID 31665279

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: CTC Retainer + Essix Retainer: The CTC is bonded directly after debonding. The Essix retainer maxilla is handed out to the patient the same day after removal of fixed appliances.
  Alginate impressions are taken at the follow-up visits. Questionnaires are completed at the follow-up visits.
  CTC retainer: The CTC retainer consists of 0.8 hard Remanium® wire (Dentaurum, Germany) and is bonded with Tetric Flow (Ivoclar Vivadent, Liechtenstein) to the lower canines directly after debonding.
  Essix retainer maxilla: The Essix retainer is made of 1 mm Essix C+® Plastic (Dentsply, USA) and is handed out to the patient the same day after removal of fixed appliances.
  Alginate impression: Alginate impressions are taken to made the cuspid-to-cuspid and Essix retainers, respectively. Dental casts are obtained at the debond appointment and at the follow-up visits after 6, 18 and 60 months.
  Questionnaire: A questionnaire is completed at the follow-up visits.
- Group B: Essix Retainer + Essix Retainer: The Essix retainer maxilla and Essix retainer mandible are handed out to the patient the same day after removal of fixed appliances.
  Alginate impressions are taken at the follow-up visits. Questionnaires are completed at the follow-up visits.
  Essix retainer maxilla: The Essix retainer is made of 1 mm Essix C+® Plastic (Dentsply, USA) and is handed out to the patient the same day after removal of fixed appliances.
  Essix retainer mandible: The Essix retainer is made of 1 mm Essix C+® Plastic (Dentsply, USA) and is handed out to the patient the same day after removal of fixed appliances.
  Alginate impression: Alginate impressions are taken to made the cuspid-to-cuspid and Essix retainers, respectively. Dental casts are obtained at the debond appointment and at the follow-up visits after 6, 18 and 60 months.
  Questionnaire: A questionnaire is completed at the follow-up visits.
Period: Overall Study
Arm/Group | Group A: CTC Retainer + Essix Retainer | Group B: Essix Retainer + Essix Retainer
Started | 52 | 52
Completed | 39 | 35
Not Completed | 13 | 17

BASELINE CHARACTERISTICS:
Population: adolescent patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: CTC Retainer + Essix Retainer | Group B: Essix Retainer + Essix Retainer | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.1 (1.9) | 17.1 (2.4) | 17.1 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 26 | 26 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 52 | 52 | 104
Region of Enrollment [Number; unit: participants]
  Sweden | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Changes in Tooth Position
Description: Analyses of changes in tooth position on dental casts Little's Irregularity Index (in mm) 0=no crowding/irregularity, higher scores= more crowding/irregularity (worse outcome)
Time Frame: Changes in tooth position (Little's Irregularity Index) were analysed 5 years (T4) after debonding (T1)
Population: Dental casts were analysed. As data were not normal distributed, median values are reported.
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Group A: CTC Retainer + Essix Retainer | Group B: Essix Retainer + Essix Retainer
Number analyzed (Participants) | 39 | 35
millimeters | 0.05 [-0.40 to 0.73] | 0.62 [-0.08 to 1.49]
Statistical Analysis 1: Comparison: Group A: CTC Retainer + Essix Retainer vs Group B: Essix Retainer + Essix Retainer; Test type: Other — GEE analysis; p = 0.0002, GEE analysis; GEE analysis = 0.99, 95% CI 2-sided [0.48 to 1.51]

2. Secondary Outcome: Patients' Perception
Description: Analyses of patients' perception by validated self-report questionnaires to evaluate experiences of the retention techniques VAS (visual analog scale, 0-100) 0= low satisfaction 100= high satisfaction
Time Frame: T4 (5 years follow up)
Population: Adolescent patients at debond (baseline), adults after 5 years
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group A: CTC Retainer + Essix Retainer | Group B: Essix Retainer + Essix Retainer
Number analyzed (Participants) | 39 | 35
score on a scale | 93 [79 to 98] | 92 [69 to 96]
Statistical Analysis 1: Comparison: Group A: CTC Retainer + Essix Retainer vs Group B: Essix Retainer + Essix Retainer; Test type: Other — Mann-Whitney U test; p = 0.55, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Observation time: 5 years after debonding (T1-T4)
Arm/Group | Group A: CTC Retainer + Essix Retainer | Group B: Essix Retainer + Essix Retainer
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-07-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT03070444/Prot_SAP_000.pdf